CLINICAL TRIAL: NCT04239118
Title: New Technologies for Endoscopic Treatment of Bleeding Gastroduodenal Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Voronezh N.N. Burdenko State Medical Academy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cherednikov
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Ulcer Hemorrhage
Keywords: ulcer; bleeding; treatment; aseptisorb-A
MeSH Terms: conditions — Ulcer; Hemorrhage | interventions — Platelet Count

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Applications of autoplasma, enriched with platelets and (Experimental): Endoscopic applications of autoplasma, enriched with platelets and granular sorbent aseptisorb-A in bleeding gastroduodenal ulcers
  Interventions: Combination Product: Complex endoscopic treatment with the use of granular sorbent aseptisorb-A and autoplasm enriched with platelets
- Traditional methods of endoscopic hemostasis (Other): Traditional methods of endoscopic hemostasis were used without the use of platelet-enriched plasma and granular sorbents.
  Interventions: Procedure: Traditional methods of endoscopic hemostasis

INTERVENTIONS:
Combination Product: Complex endoscopic treatment with the use of granular sorbent aseptisorb-A and autoplasm enriched with platelets — Complex endoscopic bleeding ulcers treatment with the use of granular sorbent aseptisorb-A and autoplasm enriched with platelets
  Arms: Applications of autoplasma, enriched with platelets and
Procedure: Traditional methods of endoscopic hemostasis — Traditional methods of endoscopic hemostasis were used without the use of platelet-enriched plasma and granular sorbents
  Arms: Traditional methods of endoscopic hemostasis

SUMMARY:
The purpose of the study was to improve treatment results of patients with bleeding gastroduodenal ulcers by endoscopic applications of autoplasma, enriched with platelets and granular sorbent aseptisorb-A.

DETAILED DESCRIPTION:
The clinical study was conducted on the basis of the Voronezh city specialized Center for the treatment of patients with gastrointestinal bleeding. The study included 112 patients with ulcerative gastroduodenal bleeding. All patients were divided into two groups by random sampling: the main group (n=57 people) and the comparison group (n=55 people). In the treatment of patients of the main group (57 people), an individual approach was used with the use of granular sorbent aseptisorb-A and autoplasm enriched with platelets, in the complex endoscopic treatment of bleeding-complicated gastroduodenal ulcers (Patent Russian Federation (RF) № 2632771). In the comparison group (55 people), traditional methods of endoscopic hemostasis were used.

ELIGIBILITY:
Inclusion Criteria:

* Gastroduodenal ulcers with bleeding

Exclusion Criteria:

* Bleedings of other etiology

Ages: 44 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
the timing of final hemostasis | a week
  the timing of final hemostasis

SECONDARY OUTCOMES:
the frequency of recurrent bleeding | 1 year
  the frequency of recurrent bleeding
mortality rates | 1 year
  mortality rates
healing of ulcerative defects | 1 year
  sizes of ulcerative defects

CONTACTS AND LOCATIONS:
Locations (1):
- Voronezh State Medical University, Voronezh, Russia

IPD SHARING:
Plan to Share IPD: No